CLINICAL TRIAL: NCT02447939
Title: A Phase I Study to Evaluate the Pharmacokinetics and Safety of Repeat Oral Doses of Dabrafenib and the Combination of Dabrafenib With Trametinib in Chinese Subjects With Melanoma
Brief Title: Pharmacokinetics of Repeat Oral Doses of Dabrafenib and the Combination of Dabrafenib and Trametinib in Chinese Subjects With Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in strategy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201020
Record Dates: First submitted 2015-05-07; First posted 2015-05-19 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: pharmacokinetics; trametinib; cutaneous melanoma; dabrafenib; safety
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib and Trametinib (Experimental): Subject will be assigned in 2 cohorts, in cohort A, subjects will be administered dabrafenib (150 mg BID) monotherapy from Day1 to Day 21 (first part), followed by dabrafenib (150 mg BID) and trametinib (2mg QD) combination (second part, starting from day 22). After the last subject in cohort A has finished the last pharmacokinetic sampling(1st part ), another 10 subjects will be enrolled in cohort B with administration of dabrafenib (150 mg BID) in combination with oral trametinib (2mg QD).
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be provided as 50 mg and 75 mg capsules. Each capsule will contain 50 mg or 75 mg of free base (present as the mesylate salt).
Drug: Trametinib — Trametinib study will be provided as 0.5 mg and 2.0 mg tablets. Each tablet will contain 0.5 mg or 2.0 mg of trametinib parent (present as the DMSO solvate)

SUMMARY:
Present clinical study will be conducted in China to evaluate the pharmacokinetics (PK) of single and repeat oral doses of dabrafenib alone and dabrafenib and trametinib in combination, the safety profile and the clinical activity of dabrafenib in combination with trametinib in Chinese melanoma subjects with BRAF V600E/K mutation. Approximately 20 evaluable subjects will be enrolled in the study, out of which, the first 10 subjects will be enrolled into cohort A (Part I and II) and remaining 10 subjects will be enrolled in cohort B. Subjects in cohort A (Part I) will receive dabrafenib 150 mg twice daily (BID) and subjects in cohort A (Part II) and Cohort B will receive combination of dabrafenib 150 mg BID and trametinib 2 mg once daily (QD). Study treatment will continue until disease progression, death or unacceptable toxicity. After disease progression, all enrolled subjects will be followed up for overall survival. The study will be completed after all subjects have died or surviving subjects have had at least 5 years of follow-up, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent.
* Males and females >=18 years of age.
* Histologically confirmed cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV (metastatic), and BRAF V600E/K mutation-positive from the designated qualified laboratory for this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate baseline organ function defined by: Absolute neutrophil count (ANC): >=1,200 /microliter (uL); Hemoglobin: >=9 grams (g)/deciliter (dL); Platelets: >=100,000 /uL; Prothrombin time/ International normalization ratio and activated partial thromboplastin time: <=1.3 x Upper Limit of Normal (ULN); Total bilirubin: <=1.5 x ULN; Aspartate aminotransferase and Alanine aminotransferase: <=2.5 x ULN; Calculated creatinine clearance (Calculate creatinine clearance using standard Cockcroft-Gault formula): >=50 milliliter (mL)/ minute (min) or 24-hour urine creatinine clearance>=50 mL/min; Left ventricular Ejection fraction (LVEF): >/= 50% LVEF in case there is no established Lower limit of normal (LLN) for a given institution.

Exclusion Criteria:

* Prior treatment with a BRAF inhibitor or a MEK inhibitor
* Pregnant or Lactating female.
* History of another malignancy. Subjects with any previous malignancy with confirmed activating RAS mutation at any time are not eligible. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility. Exception: Subjects who have been disease-free for 5 years (except those with confirmed activating RAS mutations), or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Brain metastasis are excluded unless: All known lesions have been definitively treated with surgery or stereotactic surgery (whole-brain radiation may be given as adjuvant treatment), OR Brain lesion(s), if still present, must be confirmed stable (i.e., no increase in lesion size) for >=12 weeks prior to enrollment (stability must be confirmed with two consecutive magnetic resonance image (MRI) or computed tomography (CT) scans with contrast, separated by >6 weeks AND Asymptomatic with no corticosteroid requirements for >=4 weeks prior to enrollment, AND No enzyme inducing anticonvulsants for >=2 weeks prior to enrollment. In addition, for subjects that had brain metastases but currently have no evidence of disease (NED), NED for >=12 weeks is required and must be confirmed by two consecutive scans, separated by >=6 weeks, prior to enrollment.
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to enrolment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrolment.
* Any prohibited medication(s).
* Administration of an investigational study treatment within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment(s) in this study.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* A history or evidence of cardiovascular risk including any of the following: Current LVEF < Institutional LLN; a QTc interval corrected for heart rate >=480 millisecond (msec) (using Bazett's formula); a history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with atrial fibrillation controlled for >30 days prior to enrollment are eligible; a history (within 6 months prior to enrollment) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty; a history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines; treatment refractory hypertension defined as a blood pressure of systolic>140 millimeters of mercury (mmHg) and/or diastolic >90 mm Hg which cannot be controlled by anti-hypertensive therapy; subjects with intra-cardiac defibrillators; abnormal cardiac valve morphology (>=Grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia determined by blood chemistry), long QT syndrome or taking medicinal products known to prolong the QT interval.
* A history of retinal vein occlusion (RVO)
* History of interstitial lung disease or pneumonitis.
* History of HIV infection.
* History of Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
* Subjects with laboratory evidence of cleared HBV and/or HCV will be permitted, which defined as HBs antigen negative and HBV Deoxyribonucleic acid (DNA) negative; and HCV antibody is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite of PK parameters of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) dose: Cmax,Tmax and AUC(0-tau) | At Day 1: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
  Maximum observed plasma concentration (Cmax), time to Cmax (Tmax) and area under the concentration-time curve over the dosing interval [AUC(0-tau)] will be calculated for dabrafenib and its metabolites.
A Composite of PK parameters of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) dose : Tmax, Css_min, Css_max, Css_av and AUC(0-tau) | At Day 21: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
  Tmax, minimum concentration at steady state (Css_min), maximum concentration at steady state (Css_max), average concentration at steady state (Css_av), AUC(0-tau) will be calculated for dabrafenib and its metabolites.
Accumulation ratio of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) dose | At Day 21.
Composite of PK parameters of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose: Cmax, Tmax, AUC(0-tau) | At Day 1: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
Composite of PK parameters of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose : Tmax, Css_min, Css_max, Css_av, AUC(0-tau) | At Day 21: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
Accumulation ratio of dabrafenib and its metabolites following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose | At Day 21.
Composite of PK parameters of trametinib following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose: Cmax, Tmax, AUC(0-tau) | At Day 1: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
Composite of PK parameters of trametinib following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose : Tmax, Css_min, Css_max, Css_av, AUC(0-tau) | At Day 21: Pre dose, 1,2, 3, 4, 6, 8, 12 and 24 h post dose.
Accumulation ratio of trametinib following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose | At Day 21.
Effective half-life of trametinib following single and repeat dabrafenib (150 mg BID) and trametinib (2 mg QD) dose | At Day 21.

SECONDARY OUTCOMES:
Composite of Physical examination assessment | Up to 30 days of the subject's last dose (assessed up to 5 years).
  Physical examination will include assessments of eyes, neurological and cardiovascular systems, lungs, abdomen, head, neck, ears, nose, mouth, throat, thyroid, lymph nodes, extremities, and skin, genitourinary (pelvic) and rectal exams.
Composite of Safety and tolerability as assessed by vital signs assessment: blood pressure, temperature and pulse rate | Up to 30 days of the subject's last dose (assessed up to 5 years).
  Vital sign measurements will include systolic and diastolic blood pressure, body temperature and pulse rate.
Electrocardiogram (ECG) assessment | Up to 30 days of the subject's last dose (assessed up to 5 years).
  12-lead ECGs will be obtained at each time point using an ECG machine that automatically to calculate the heart rate and measures PR, QRS, QT and corrected QT interval duration (QTc intervals).
Echocardiogram (ECHO) assessment | At week 4, week 8, and then every 8 weeks until treatment discontinuation.
  ECHO assessment will include an evaluation for left ventricular ejection fraction.
Eye exams assessment | At screening, and when clinical indicated until treatment discontinuation.
  Eye exam will include indirect fundoscopic examination,visual acuity, visual field examination, and tonometry, with special attention to retinal abnormalities.
Chemistry laboratory values assessment | Up to 30 days of the subject's last dose (assessed up to 5 years).
Number of subjects with Adverse events (AEs) | Up to 5 years.
Number of subjects with Serious Adverse events (SAEs) | Up to 5 years.
Objective response rate (ORR) | Up to 5 years.
  ORR defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation
Progression free survival(PFS) | Up to 5 years.
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Overall survival(OS) | Up to 5 years.
  OS defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact.
Hematology laboratory values assessment | Up to 30 days of the subject's last dose (assessed up to 5 years).
Urinalysis laboratory values assessment | Up to 30 days of the subject's last dose (assessed up to 5 years).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline